CLINICAL TRIAL: NCT07062068
Title: Comparative Study Between Ultrasound-Guided Brachiocephalic Vein and Internal Jugular Vein Cannulation in Mechanically Ventilated ICU Patients
Brief Title: Ultrasound-Guided BCV and IJV in ICU Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hasnaa Mohy Ibrhim, Resident doctor at department of anesthesia and ICU, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SU-BCV-IJV-2025
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Ultrasound-Guided Vascular Access; ICU Patients
Keywords: Comparative Study Between Ultrasound-Guided Brachiocephalic Vein and Internal Jugular Vein Cannulation in Mechanically Ventilated ICU Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- candidates for BCV cannulation (Active Comparator)
  Interventions: Procedure: ultrasound guided Brachiocephalic vein and internal jugular vein cannulation in mechanically ventilated ICU patients
- candidates for IJV cannulation (Active Comparator)
  Interventions: Procedure: ultrasound guided Brachiocephalic vein and internal jugular vein cannulation in mechanically ventilated ICU patients

INTERVENTIONS:
Procedure: ultrasound guided Brachiocephalic vein and internal jugular vein cannulation in mechanically ventilated ICU patients — For Arm ( candidates for BCV cannulation ) :
  by ultrasound guided we insert Central venous catheter in BCV under complete aseptic condition For Arm ( candidates for IJV cannulation ) by ultrasound guided we insert central venous catheter in IJV under complete aseptic conidtion we do comparison between the 2 arms as regard : 1st pass success rate , complications and failure rate in ventilated patient in ICU .

SUMMARY:
This is a prospective randomized clinical trial aiming to compare the success rate, complications, and insertion time between ultrasound-guided brachiocephalic vein (BCV) and internal jugular vein (IJV) cannulation in mechanically ventilated patients in the intensive care unit (ICU). The goal is to determine whether BCV access offers a safer or more effective alternative in critically ill patients requiring central venous catheter placement.

DETAILED DESCRIPTION:
Central venous cannulation is a common and essential procedure in the management of critically ill patients, especially those requiring mechanical ventilation. Traditionally, the internal jugular vein (IJV) has been the preferred site. However, the brachiocephalic vein (BCV) has recently gained attention due to its potentially favorable anatomical location and reduced complication rates.

This study is designed to compare the outcomes of ultrasound-guided cannulation of the BCV versus the IJV, focusing on parameters such as success rate of insertion on first attempt, total cannulation time, and incidence of complications such as arterial puncture, pneumothorax, or hematoma formation. The study will be conducted on adult patients admitted to the ICU and undergoing mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

100 patients with age between ( 18 - 50 years old ) ventilated in ICU with need central venous access , with physical status II or III according to ASA classification .

Exclusion Criteria:

* refusal of relatives of patients
* Any contraindication of Central venous line insertion as thrombocytopenia , coagulopathy …. Etc
* any suspected or documented thrombus inside vein
* any congenital or acquired musculo-skeletal deformities of neck or clavicle
* any active infections or signs of inflammation over insertion site
* any previous procedures performed at the cannulation site

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
cannulation failure rate | Baseline
  Failure to cannulate selected vein at 1st attempt

IPD SHARING:
Plan to Share IPD: Undecided